CLINICAL TRIAL: NCT03661073
Title: Comprehensive Assessment of Motor Imagery Ability After Stroke
Brief Title: Motor Imagery Ability After Stroke
Acronym: AVCIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL18_0059
Record Dates: First submitted 2018-06-01; First posted 2018-09-07 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke (Experimental): The investigator will include patients with stroke (either hemorrhagic or ischemic) with or without neglect in the experimental group.
  Interventions: Behavioral: Assessment of motor imagery ability
- Healthy subjects (Sham Comparator): The investigator will include healthy subjects aged-matched to participants of the experimental group in the control group.
  Interventions: Behavioral: Assessment of motor imagery ability of healthy subject

INTERVENTIONS:
Behavioral: Assessment of motor imagery ability — The intervention will last 3 hours ± 45 minutes, the assessment will be spread over 3 sessions of 1 hour ± 15 minutes on one week. The time between two sessions will depend on patient fatigability and availability. The VMIQ-2 and the KVIQ-20 will be realized during the first session. In the second session, patients will perform the hand laterality judgment task and the MIQ-RS. During the last session the Timed up and go and the box and block test will be realized.
  Arms: Stroke
Behavioral: Assessment of motor imagery ability of healthy subject — The intervention will last 2 hours ± 15 minutes. All the tests will be spread over 1 session. Assessment order will be VMIQ-2, KVIQ-20, the hand laterality judgment task, the after a break MIQ-RS, iTUG and iBBT.
  Arms: Healthy subjects

SUMMARY:
Individuals with stroke may experience sensory-motor deficit and/or neglect, with possible reduction in motor imagery ability (MI). To our knowledge, no study completely investigated MI ability in one individual whereas MI practice can be performed using visual or kinesthetic modalities (respectively visualizing with mind's eyes or imagining movement using sensation) and internal or external perspectives (performing action as spectator or as actor). This study aims to investigate MI ability in patients with stroke as compared to aged-matched healthy individuals. The investigators will assess explicit MI ability using 3 questionnaires (Movement Imagery Questionnaire-RS - MIQ-RS, Kinesthetic and Visual Imagery Questionnaire-20 - KVIQ-20, Vividness of Movement Imagery Questionnaire-2 - VMIQ-2) and 2 tests (imagined Time Up and Go - iTUG, imagined Box and Block test - iBBT). Outcome parameters will be i) the composite score of vividness measured for all tests using Likert scales, ii) the temporal equivalence between MI and Physical practice (PP - where MI/PP ratio equal to 1 indicate good MI ability and respect of temporal equivalence between MI and PP) and iii) the amplitude of electrodermal activity. The investigators will also study implicit MI ability using a hand laterality judgment task. Outcomes parameters will be response time (i.e. the duration to identify the hand laterality) and the percentage of correct responses.

ELIGIBILITY:
Inclusion Criteria:

For both groups:

* be more than 18 years old
* be less than 75 years old
* benefit from social security

For experimental group:

* patient admitted in Henry Gabrielle hospital for rehabilitation
* patient with one single episode of stroke

Exclusion Criteria:

For patients:

* sign of cognitive decline (MMSE score under 27/30)
* evolutionary pathology associated

For healthy subjects:

- neurological or orthopaedical history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Score of vividness | Day 1
  Participants will self-report vividness that describe the success in imagining movements using a 5-points Likert scale (1=no image or no sensation to 5=image as clear as PP or sensation as intense as PP) for the KVIQ-20. The investigators will average the vividness for each items of the questionnaire.

SECONDARY OUTCOMES:
Temporal equivalence measured during KVIQ-20 | Day 1
  The investigators will time the duration of physical practice (PP) and motor imagery (MI) movements, and then compute a ratio MI/PP for each item and average these ratios to get a measure of temporal equivalence for the KVIQ-20.
Amplitude of electrodermal responses that will be measured during imagined movement with reference to actual movements measured during KVIQ-20. | Day 1
  The investigators will measure amplitude of electrodermal response during actual and imagined movement. The investigators will average the amplitude of response and compute the ratio imagined/actual expressed in percent for the KVIQ-20.
Score of vividness measured during VMIQ -2 | Day 1
  Participants will self-report vividness that describe the success in imagining movements using a 5-points Likert scale (1=no image or no sensation to 5=image as clear as PP or sensation as intense as PP) for the VMIQ -2. The investigators will average the vividness for each items of the questionnaire.
Amplitude of electrodermal responses that will be measured during imagined movement with reference to actual movements measured during VMIQ -2. | Day 1
  The investigators will measure amplitude of electrodermal response during actual and imagined movement. The investigators will average the amplitude of response and compute the ratio imagined/actual expressed in percent for the VMIQ -2.
Score of vividness measured during MIQ-RS. | Day 3
  Participants will self-report vividness that describe the success in imagining movements using a 7-points Likert scale a 7-points Likert scale for MIQ (1=very difficult to imagine to 7=very easy to imagine) for the VMIQ -2. The investigators will average the vividness for each items of the questionnaire.
Temporal equivalence measured during MIQ-RS. | Day 3
  The investigators will time the duration of physical practice (PP) and motor imagery (MI) movements. Then the investigators will compute a ratio MI/PP for each item and average these ratios to get a measure of temporal equivalence for the MIQ-RS.
Amplitude of electrodermal responses that will be measured during imagined movement with reference to actual movements measured during MIQ-RS. | Day 3
  The investigators will measure amplitude of electrodermal response during actual and imagined movement. The investigators will average the amplitude of response and compute the ratio imagined/actual expressed in percent for the MIQ-RS.
Percentage of correct response to identify the hand laterality during the implicit motor imagery ability assessment | Day 3
  Participant will have to identify the hand laterality of the 196 hand pictures successively displayed on a computer screen with different rotation and orientation (namely palm, back, thumb, pinky). The investigators will record the response and compute the averaged percentage of correct response.
Response time to identify the hand laterality during the implicit motor imagery ability assessment | Day 3
  Participant will have to identify the hand laterality of the 196 hand pictures successively displayed on a computer screen with different rotation and orientation (namely palm, back, thumb, pinky). The investigators will time the duration to indicate the response and compute the averaged the response time for identification.
Score of vividness measured during iTUG. | Day 5
  Participants will self-report vividness that describe the success in imagining movements using a 5-points Likert scale (1=no image or no sensation to 5=image as clear as PP or sensation as intense as PP) for the iTUG. The investigators will average the vividness for each items of the questionnaire.
Temporal equivalence measured during iTUG. | Day 5
  The investigators will time the duration of physical practice and motor imagery movements three consecutive times. Then the investigators will compute a ratio MI/PP for time and average these ratios to get a measure of temporal equivalence for the iTUG.
Amplitude of electrodermal responses that will be measured during imagined movement with reference to actual movements measured during iTUG. | Day 5
  The investigators will measure amplitude of electrodermal response during actual and imagined movement. The investigators will average the amplitude of response and compute the ratio imagined/actual expressed in percent for the iTUG.
Score of vividness measured during iBBT. | Day 5
  Participants will self-report vividness that describe the success in imagining movements using a 5-points Likert scale (1=no image or no sensation to 5=image as clear as PP or sensation as intense as PP) for the iBBT. The investigators will average the vividness for each items of the questionnaire.
Temporal equivalence measured during iBBT. | Day 5
  The investigators will time the duration of physical practice and motor imagery movements three consecutive times. Then the investigators will compute a ratio MI/PP for time and average these ratios to get a measure of temporal equivalence for the iBBT.
Amplitude of electrodermal responses that will be measured during imagined movement with reference to actual movements measured during iBBT. | Day 5
  The investigators will measure amplitude of electrodermal response during actual and imagined movement. The investigators will average the amplitude of response and compute the ratio imagined/actual expressed in percent for the iBBT.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henry Gabrielle, Saint-Genis-Laval, France